CLINICAL TRIAL: NCT00385632
Title: Quality of Life and Healthcare Utilization Substudy
Brief Title: Effects of Two Anti-HIV Drug Regimens on Quality of Life and Health Care Use Among SMART Study Participants
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Community Programs for Clinical Research on AIDS (Network)
Responsible Party: Sponsor
Other Study IDs: CPCRA 065A; SMART; 10112 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Participants following a drug conservation (DC) regimen in which ART was stopped or deferred until CD4 cell count dropped below 250 cells/mm3, initiated until CD4 cell count was at least 350 cells/mm3, and then followed by episodic ART based on CD4 cell count
  Interventions: Drug: Antiretroviral Regimens
- 2: Participants following a viral suppression (VS) regimen in which ART was continued to keep viral loads as low as possible, regardless of CD4 cell count
  Interventions: Drug: Antiretroviral Regimens

INTERVENTIONS:
Drug: Antiretroviral Regimens — Various antiretroviral therapy combinations already being administered to participants

SUMMARY:
The purpose of this study is to compare the effects of two different anti-HIV drug regimens on quality of life and health care utilization among SMART study participants.

DETAILED DESCRIPTION:
Advances in antiretroviral therapy (ART) have dramatically reduced mortality and morbidity rates for HIV infected people. However, HIV infection is a costly disease to treat. With improvement in survival, quality of life and the long-term cost of HIV treatment have become increasingly important to the majority of individuals infected with HIV. Different HIV treatment regimens may lead to variations in quality of life and health care costs over the course of treatment. In the SMART study, participants were randomly assigned to one of two treatment groups:

* Group 1 participants followed a drug conservation (DC) regimen in which ART was stopped or deferred until CD4 cell count dropped below 250 cells/mm3, initiated until CD4 cell count was at least 350 cells/mm3, and then followed by episodic ART based on CD4 cell count.
* Group 2 participants followed a viral suppression (VS) regimen in which ART was continued to keep viral loads as low as possible, regardless of CD4 cell count.

The purpose of this study is to compare how the DC and VS regimens affect quality of life, symptom severity, health care utilization, and resulting costs among SMART study participants.

At baseline, participants will complete questionnaires regarding quality of life, symptoms, health care utilization, current insurance, and socioeconomic status. Body appearance and signs of HIV disease progression will also be assessed at this time. Follow-up evaluations on quality of life and symptoms will be repeated at Months 4, 8, and 12 and annually thereafter. Follow-up evaluations of all other baseline measures will occur once a year.

ELIGIBILITY:
Inclusion Criteria:

* Coenrollment in the SMART study
* Parent or guardian willing to provide informed consent, if applicable

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants using conservation and viral suppression ART treatment regimens
Sampling Method: Non-Probability Sample
Enrollment: 1224 (Actual)
Dates: Start 2002-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Quality of life as assessed by self-administered questionnaires, a symptom severity survey, and an assessment of body appearance | Throughout study
Self-reported healthcare utilization | Throughout study
Recorded medications used by participants | Throughout study
Cost of treating HIV/AIDS | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, MD, MPH, Study Chair — Harlem AIDS Treatment Group, Harlem Hospital Center; James Neaton, PhD, Study Chair — CPCRA Statistical and Data Management Center/CCBR
Locations (67):
- United States (67):
  - UCSF, Fresno, School of Medicine, Dept. of Internal Medicine CRS, Fresno, California
  - Dr. M. Estes Med. Practice CRS, Mill Valley, California
  - Dr. Robert Scott Med. Practice CRS, Oakland, California
  - East Bay AIDS Ctr. CRS, Oakland, California
  - Dr. Shawn Hassler Med. Practice CRS, San Francisco, California
  - Positive Health Program Clinic (San Francisco Gen. Hosp.) CRS, San Francisco, California
  - Dr. Virginia Cafaro Med. Practice CRS, San Francisco, California
  - Dr. William Owen Med. Practice CRS, San Francisco, California
  - Castro-Mission Health Ctr. CRS, San Francisco, California
  - San Francisco VAMC, Infectious Diseases Clinic CRS, San Francisco, California
  - UCSF PHP, Gen. Internal Medicine Practice CRS, San Francisco, California
  - Beacon Clinic at Boulder CRS, Boulder, Colorado
  - Denver Infectious Diseases Consultants CRS, Denver, Colorado
  - Kaiser Permanente of Denver CRS, Denver, Colorado
  - Univ. of Colorado Health Science Ctr. CRS, Denver, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Eastside Family Health Ctr. CRS, Denver, Colorado
  - Denver VAMC CRS, Denver, Colorado
  - Denver Public Health CRS - INSIGHT, Denver, Colorado
  - Western Infectious Disease Consultants CRS, Wheat Ridge, Colorado
  - Univ. of Connecticut Health Ctr. CRS, Farmington, Connecticut
  - Yale Univ. School of Medicine, NE ProACT - New Haven CRS, New Haven, Connecticut
  - Hosp. of St. Raphael CRS, New Haven, Connecticut
  - VAMC West Haven CRS, West Haven, Connecticut
  - Georgetown Wellness Clinic, Georgetown, Delaware
  - Christiana Care Health Services HIV Program CRS, Wilmington, Delaware
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - Miami VAMC CRS, Miami, Florida
  - Atlanta VAMC CRS, Decatur, Georgia
  - Klein & Slotten Medical Associates CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Univ. of Illinois Family Ctr. for Infectious Disease CRS, Chicago, Illinois
  - Univ. of Chicago Hosps. CRS, Chicago, Illinois
  - Lakeshore Infectious Disease Associates CRS, Chicago, Illinois
  - North Side Family Medicine CRS, Chicago, Illinois
  - Northwestern Memorial Physicians Group CRS, Chicago, Illinois
  - Earl K. Long Med. Ctr., LSU - Mid City EIC Clinic CRS, Baton Rouge, Louisiana
  - James Osterberger, MD (Private Med. Practice) CRS, Baton Rouge, Louisiana
  - Med. Ctr. of Louisiana at New Orleans, HIV Outpatient Clinics CRS, New Orleans, Louisiana
  - Tulane University Health Sciences Center, Louisiana Community AIDS Research Program(LaCARP) CRS, New Orleans, Louisiana
  - New Orleans VAMC CRS, New Orleans, Louisiana
  - CRI-Boston CRS, Boston, Massachusetts
  - CRI-Springfield CRS, Springfield, Massachusetts
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Univ. of Mississippi Med. Ctr., Div. of Infectious Diseases CRS, Jackson, Michigan
  - Michigan State Univ., Infectious Disease Clinic CRS, Lansing, Michigan
  - Mt. Clemens Gen. Hosp. CRS, Mount Clemens, Michigan
  - Providence Hosp,-Newland Med. Assoc Inc CRS, Southfield, Michigan
  - ID Care Inc. - Hillsborough CRS, Hillsborough, New Jersey
  - Cathedral Healthcare System, St. Michael's Med. Ctr. CRS, Newark, New Jersey
  - New Jersey Community Research Initiative, Jeffrey Bomser Clinic CRS, Newark, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey CRS, Paterson, New Jersey
  - Raritan Bay Med. Ctr., Perth Amboy Division CRS, Perth Amboy, New Jersey
  - ID Care - Randolph CRS, Randolph Township, New Jersey
  - Infectious Disease Specialists of N.J., North Jersey Community Research Initiative CRS, Union, New Jersey
  - St. Vincent Hosp. & Med. Ctr. CRS, New York, New York
  - Metropolitan Hosp. Ctr. CRS, New York, New York
  - Harlem Hospital Ctr./Columbia University CRS (Gordin CTU), New York, New York
  - Harlem Hosp. Ctr., Outpatient Clinics (New York) CRS, New York, New York
  - Jacobi Med. Ctr., Ambulatory Care Pavillion CRS, The Bronx, New York
  - Legacy Community Health Services, Inc. CRS, Houston, Texas
  - Baylor College of Medicine, Thomas St. Clinic CRS, Houston, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Michael E. DeBakey VAMC CRS, Houston, Texas
  - Thomas Street Clinic CRS, Houston, Texas
  - Univ. Clinical Research Ctr., Memorial Hermann Hosp. CRS, Houston, Texas
  - South Texas Veterans Health Care System, Immunosuppression Clinic CRS, San Antonio, Texas

REFERENCES:
- [Background] Anis AH, Guh D, Hogg RS, Wang XH, Yip B, Craib KJ, O'Shaughnessy MV, Schechter MT, Montaner JS. The cost effectiveness of antiretroviral regimens for the treatment of HIV/AIDS. Pharmacoeconomics. 2000 Oct;18(4):393-404. doi: 10.2165/00019053-200018040-00007. PMID 15344307
- [Background] Byrne MW, Honig J. Health-related quality of life of HIV-infected children on complex antiretroviral therapy at home. J Assoc Nurses AIDS Care. 2006 Mar-Apr;17(2):27-35. doi: 10.1016/j.jana.2006.01.003. PMID 16800165
- [Background] Liu C, Ostrow D, Detels R, Hu Z, Johnson L, Kingsley L, Jacobson LP. Impacts of HIV infection and HAART use on quality of life. Qual Life Res. 2006 Aug;15(6):941-9. doi: 10.1007/s11136-005-5913-x. PMID 16900275
- [Background] Lowy A, Page J, Jaccard R, Ledergerber B, Somaini B, Weber R, Szucs T. Costs of treatment of Swiss patients with HIV on antiretroviral therapy in hospital-based and general practice-based care: a prospective cohort study. AIDS Care. 2005 Aug;17(6):698-710. doi: 10.1080/09540120412331336689. PMID 16036256
- See also: Click here for more information on CPCRA 065 — http://clinicaltrials.gov/show/NCT00027352